CLINICAL TRIAL: NCT04287478
Title: A Phase I/II Study of Bacteriophage Therapy to Evaluate Safety, Tolerability, and Efficacy of Targeted "Personalized" Bacteriophage Treatments in Patients With Bacterial Infection of the Urinary Tract
Brief Title: Bacteriophage Therapy in Patients With Urinary Tract Infections
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to a change in development strategy.
Sponsor: Adaptive Phage Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APT.UTI.001
Record Dates: First submitted 2020-02-03; First posted 2020-02-27 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infection Bacterial
Keywords: Antimicrobial Resistance; Bacteriophage; Urinary Tract Infections; Phage
MeSH Terms: conditions — Urinary Tract Infections | interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Initially, patients with neurogenic bladder and urinary tract infections will be enrolled and followed for bacterial eradication. Results from this cohort will be used to confirm or modify the phage dosing regimen before proceeding to the patients with symptomatic infection at risk of recurrence. The trial will use pre-specified criteria to determine what phage regimens should be evaluated.
Masking Description: Patient will be randomized to receive either active phage or placebo treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Intravenous (IV) (Experimental): Phage administered via the intravenous route.
  Interventions: Biological: Bacteriophage Therapy
- Intravesical (IVS) (Experimental): Phage administered via the intravesical route.
  Interventions: Biological: Bacteriophage Therapy
- Subcohort A (Experimental): Selected phage for E. coli administered via selected route based on previous Arms.
  Interventions: Biological: Bacteriophage Therapy
- Subcohort B (Experimental): Selected phage for Klebsiella pneumoniae administered via selected route based on previous Arms.
  Interventions: Biological: Bacteriophage Therapy
- Subcohort C (Experimental): Selected phage for E. coli administered via selected route based on previous Arms.
  Interventions: Biological: Bacteriophage Therapy
- Subcohort D (Experimental): Selected phage for Klebsiella pneumoniae administered via selected route based on previous arms.
  Interventions: Biological: Bacteriophage Therapy

INTERVENTIONS:
Biological: Bacteriophage Therapy — Bacteriophage therapy will be personalized for each patient dependent on phage susceptibility testing

SUMMARY:
This is a phase I/II trial designed to evaluate bacteriophage therapy in patients with urinary tract infections.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of bacteriophage therapy in patients with urinary tract infection (UTI). Patients to be enrolled will have urinary tract infections due to E. coli and K. pneumoniae. This will include asymptomatic patients with neurogenic bladder and symptomatic patients with complicated urinary tract infections who are at risk of UTI recurrence. Patients will be followed for bacterial clearance or recurrence of urinary tract infection.

ELIGIBILITY:
General Inclusion Criteria:

* Males or females ≥18 years of age.
* Female patients of childbearing potential.
* Male patients must agree not to donate sperm up for one month.
* English-speaking.

General Exclusion Criteria:

* Stage 4 or greater chronic kidney disease (CKD).
* Abnormal liver function tests >3×upper limit of normal (ULN).
* Other conditions which could confound study results.
* Body mass index of > 40 or weight less than 50 kg.
* Known allergy to phage products.
* Pregnant and/or breastfeeding.
* Immunocompromised.
* Need for antiviral medication.
* History of severe autonomic dysreflexia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Identify ideal bacteriophage treatment regimens based on improvements in disease control rates | baseline
  Microbiological eradication of target pathogen identified at baseline

SECONDARY OUTCOMES:
Assess the safety of bacteriophage therapy | At least 56 days
  Safety will be measured by the number and percent of treatment related adverse events.
Assess the tolerability of bacteriophage therapy | At least 56 days
  Tolerability will be measured by the percentage of patients who discontinue treatment due to adverse events

OTHER OUTCOMES:
Recurrence of urinary tract infection | 1 year
  Recurrence of urinary tract infection for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hopkins, MD, Principal Investigator — Chief Medical Officer
Locations (8):
- United States (8):
  - Universal Axon Clinical Research, Doral, Florida
  - AdMed Research, Miami, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Innovation Medical Research Center, Inc, Palmetto Bay, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - James J. Peters VA Medical Center, The Bronx, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - DHR Health Institute for Research and Development, Edinburg, Texas